CLINICAL TRIAL: NCT06132152
Title: Evaluation of Hemorrhoidectomy Techniques: Scalpel and Electrosurgery
Brief Title: Hemorrhoids: Options of Traditional Hemorrhoidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Center of Endourology "Endocenter" (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 59954654
Record Dates: First submitted 2023-11-05; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Hemorrhoids; Open Hemorrhoidectomy
Keywords: symptomatic hemorrhoids; open hemorrhoidectomy; postoperative pain; electrosurgery
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative; Hyperthermia

STUDY DESIGN:
Intervention Model Description: In case of meeting inclusion criteria of patient the selection of the group will be determined by randomization, so both groups will be recruited simultaneously
Who Masked: Participant, Outcomes Assessor
Masking Description: Before the operation, all patients are scheduled to perform an open hemorrhoidectomy, which includes radial skin-mucosal excision of enlarged hemorrhoids with ligation of the vascular pedicle. Patients are not informed about which instrument will be used.
  All collected information will be stored in electronic databases, where patient names and group numbers are anonymized and encrypted. Thus, during the statistical calculation, a person will not know about the name of the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open hemorrhoidectomy with 'cold' scalpel (Active Comparator): Open hemorrhoidectomy will be performed in traditional way, including radial skin-mucosal excision of enlarged hemorrhoids with ligation of the vascular pedicle. 'Cold' scalpel will be used for cutting the perianal skin and anal mucose. To stop and prevent bleeding the monopolar coagulation may be used but on low energy level and with no touching the skin and mucose.
  Interventions: Procedure: Open hemorrhoidectomy with 'cold' scalpel
- Open hemorrhoidectomy with electrosurgical scalpel (Active Comparator): Open hemorrhoidectomy will be performed in traditional way, including radial skin-mucosal excision of enlarged hemorrhoids with ligation of the vascular pedicle. Electrosurgical scalpel will be used during all steps including cutting the perianal skin and anal mucose and to stop and prevent bleeding.
  Interventions: Procedure: Open hemorrhoidectomy with electrosurgical scalpel

INTERVENTIONS:
Procedure: Open hemorrhoidectomy with 'cold' scalpel — Open hemorrhoidectomy will be performed in traditional way, including radial skin-mucosal excision of enlarged hemorrhoids with ligation of the vascular pedicle. 'Cold' scalpel will be used for cutting the perianal skin and anal mucose. To stop and prevent bleeding the monopolar coagulation may be used but on low energy level and with no touching the skin and mucose.
  Arms: Open hemorrhoidectomy with 'cold' scalpel
Procedure: Open hemorrhoidectomy with electrosurgical scalpel — Open hemorrhoidectomy will be performed in traditional way, including radial skin-mucosal excision of enlarged hemorrhoids with ligation of the vascular pedicle. Electrosurgical scalpel will be used during all steps including cutting the perianal skin and anal mucose and to stop and prevent bleeding.
  Arms: Open hemorrhoidectomy with electrosurgical scalpel

SUMMARY:
The goal of this prospective clinical trial is to compare the outcomes of several technical options of open hemorrhoidectomy in patients with symptomatic hemorrhoids. Randomly allocated participants will undergo surgical treatment for hemorrhoids with one technical option of open hemorrhoidecomy: with 'cold' scalpel or electrosurgical instruments. All information to evaluate outcomes between the groups will be collected before surgery and 1 week and 30 days after surgery.

DETAILED DESCRIPTION:
This is a single-center prospective randomized controlled study will be conducted on the basis of the surgical department. Patients with symptomatic hemorrhoids and who will be intended for surgical treatment (open hemorrhoidectomy) will be randomly allocated to one of the group. Prior to surgery the demographic and clinical data will be collected. Open hemorrhoidectomy under spinal anesthesia will be performed with one of the technical options according to the patient's group:

* hemorrhoidectomy with 'cold' scalpel for cutting the perianal skin and anal mucose
* hemorrhoidectomy with electrosurgical scalpel for cutting the perianal skin and anal mucose.

Intraoperative and postoperative data will be collected during first week after surgery and 30 days after surgery. Then the primary and secondary outcomes are evaluated between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Diagnosed symptomatic hemorrhoidal disease
* Planned surgery - open hemorrhoidectomy
* Absence of other anarectal diseases
* I, II class of anesthetic risk according to ASA classification
* Voluntary signing by the participant of an informed consent for surgical treatment and participation in a clinical trial.

Exclusion Criteria:

* Chronic or prolonged use of medications, including narcotic drugs, with analgesic effect for other diseases.
* Patients who have contraindications or technical impossibility of performing subarachnoid anesthesia or the full standard volume of surgery for the corresponding disease.
* Patients who refused to participate at any time before the end of the study, as well as patients who did not pass the final postoperative monitoring (1 month after the intervention).
* Pregnant women
* Complicated course of the postoperative period due to exacerbation of concomitant diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain at rest and during defecation | during 10 days after surgery
  The pain was assessed using a visual analogue scale (VAS uses a 10 cm line with endpoint descriptors such as 'no pain' marked at the left end of the line and 'worst pain imaginable' marked at the right end)

SECONDARY OUTCOMES:
Rate of prescribing opioid analgesics | 3 days after surgery
  the rate of prescribing opioid analgesics to prevent the pain from rising above VAS 5 after surgery (VAS uses a 10 cm line with endpoint descriptors such as 'no pain' marked at the left end of the line and 'worst pain imaginable' marked at the right end)
Other medications use | 10 days after surgery
  The frequency of other analgesics taken
Readmission rate | 30 days after surgery
  The number of cases of repeated appeals for relapse of the disease or hospitalizations
The life quality rate | 7 and 30 days
  The overall quality of life was assessed using the EQ-5D patient questionnaire. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
Complication rate | within 30 days after surgery
  Cases of bleeding, urinary retention, infectious complications after surgery
Residual symptoms | 30 days after surgery
  The presence of residual symptoms after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Surgical department of the Medical Research and Educational Center of Lomonosov Moscow State University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No